CLINICAL TRIAL: NCT01424787
Title: Non-interventional Study to Evaluate the Ease of Reaching Individual Goals in Serum Phosphorus (Steering)
Acronym: Steering
Status: Completed | Type: Observational
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Collaborators: Siro Clinpharm Germany GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RP-OSV-01-EU
Record Dates: First submitted 2011-08-26; First posted 2011-08-29 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2015-03

CONDITIONS: Hyperphosphataemia; ESRD
MeSH Terms: conditions — Hyperphosphatemia; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- OsvaRen treatment: Dialysis patients on OsvaRen treatment

SUMMARY:
The objective of this non-interventional study is to confirm that with standard OsvaRen® treatment it is possible to achieve in at least 60% of the patients the levels of phosphorus, total calcium, and iPTH seen in the CALMAG study also in the normal clinical practice.

DETAILED DESCRIPTION:
Only a small fraction of haemodialysis patients meet the published NKF-KDOQI standards for calcium, phosphorus, calcium x phosphorus product and intact parathyroid hormone. One of the reasons is the still difficult and insufficient therapy with phosphate binders. Even though calcium containing phosphate binders have been proven to be effective, they are reported to lead in certain patients to hypercalcaemia. This observational study therefore not only evaluates the efficacy of the phosphate binder OsvaRen® (containing calcium acetate and magnesium carbonate) but also the frequency of untoward events in daily practice as well as to the state of hyper-/ hypoparathyroidism as represented by serum iPTH values and the practice patterns used to adjust to and to fully exploit the qualities of the different available phosphate binders. In addition, the compensatory actions of the physicians, such as adaptation of the dialysate calcium or the combination with non-calcium containing phosphate binders, are going to be monitored. In order to receive additional safety data in the context of daily practice, the frequency of untoward events related to the treatment will be documented and analysed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed Informed Consent
* Patient on maintenance haemodialysis, online haemodiafiltration, or peritoneal dialysis at the time of OsvaRen® prescription
* Patients being treated with OsvaRen® for up to 6 months at the day of inclusion

Exclusion Criteria:

* Prior participation in this observational study
* Use of OsvaRen® for purposes other than those indicated in the Summary of Product Characteristics (SmPC) / package leaflet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dialysis patients (HD, HDF, or PD) being treated with OsvaRen for hyperphosphataemia
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2011-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus | 12 months

SECONDARY OUTCOMES:
Adverse drug reactions | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Geiger, MD, Prof, Principal Investigator — University Hospital, Frankfurt, Germany
Locations (24):
- Denmark (4):
  - Regionshospitalet Holstebro, Holstebro, Holstebro
  - Nykøbing Falster Sygehus, Nykøbing Mors, Nykobing
  - Roskilde Sygehus, Roskilde, Roskilde
  - Viborg Sygehus, Viborg, Viborg
- Germany (14):
  - Dialysezentrum, Aachen
  - Dialysezentrum, Alsfeld
  - Dialyszentrum/Gemeinschaftspraxis, Augsburg
  - Nephrologicum Lausitz, Cottbus
  - Studienzentrum Karlstraße, Düsseldorf
  - Dialyse am Lichtbogen, Essen
  - Diakonissenkrankenhaus Flensburg, Flensburg
  - PHV-Dialysezentrum Goslar, Goslar
  - Zentrum für Nieren-, Hochdruck- und Stoffwechselerkrankungen, Hanover
  - Gemeinschaftspraxis Nephrologie/Dialyse, Hoyerswerda
  - Internistische Schwerpunktpraxis Gastroenterologie / Nephrologie, Kaiserslautern
  - PHV Dialysezentrum Kiel, Kiel
  - Gemeinschaftspraxis Dialyse, Magdeburg
  - Dialysezentrum Pforzheim, Pforzheim
- Spain (3):
  - Hospital Infanta Leonor, Madrid
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Universitario Marqués de Valdecilla, Santander
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Western Health and Social Care Trust, Londonderry
  - Royal Shrewsbury Hospital, Shrewsbury

REFERENCES:
- [Background] de Francisco AL, Leidig M, Covic AC, Ketteler M, Benedyk-Lorens E, Mircescu GM, Scholz C, Ponce P, Passlick-Deetjen J. Evaluation of calcium acetate/magnesium carbonate as a phosphate binder compared with sevelamer hydrochloride in haemodialysis patients: a controlled randomized study (CALMAG study) assessing efficacy and tolerability. Nephrol Dial Transplant. 2010 Nov;25(11):3707-17. doi: 10.1093/ndt/gfq292. Epub 2010 Jun 7. PMID 20530499